CLINICAL TRIAL: NCT06474650
Title: A Randomized, Open-label, Two-period, Double-crossover Phase 1 Study to Evaluate the Effect of Food on the Pharmacokinetics of LPM3770164 Sustained-release Tablets in Healthy Subjects
Brief Title: Effect of Food on the Pharmacokinetics of LPM3770164 Sustained-release Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY03015/CT-CHN-103
Record Dates: First submitted 2024-06-20; First posted 2024-06-25 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Huntington Disease; Tardive Dyskinesia
MeSH Terms: conditions — Huntington Disease; Tardive Dyskinesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fed condition (Experimental): Period in which subjects receive a single oral dose of LPM3770164 sustained-release tablets in fed condition
  Interventions: Drug: LPM3770164 sustained release tablet
- Fasted condition (Experimental): Period in which subjects receive a single oral dose of LPM3770164 sustained-release tablets in fasted condition
  Interventions: Drug: LPM3770164 sustained release tablet

INTERVENTIONS:
Drug: LPM3770164 sustained release tablet — Single-dose of 30 mg of LPM3770164 sustained release tablet
  Other Names: LY03015

SUMMARY:
This is a A single-center, randomized, open-label, two-dose, two-period, crossover trial was conducted to evaluate the effect of food on the Pharmacokinetic characteristics and safety of oral administration of LPM3770164 sustained-release tablets 30 mg in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who voluntarily participate and sign the informed consent form;
2. Healthy male/female volunteers aged 18 to 45 years;
3. Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) 18.5 ~ 26.0 kg/m2, inclusive;
4. Able to comply with the lifestyle restrictions.

Exclusion Criteria:

1. Subject has a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution;
2. Subject has a current or past medical history that may affect the clinical trial or dysfunction, including but not limited to the past or current respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, motor system, blood system, psychiatry/ psychology, dermatology and other clinically serious diseases or chronic diseases; or any other diseases that may interfere with the test results;
3. Any surgical condition or condition may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects;.
4. Subject has a history of self-mutilation; or at risk of suicide;
5. Subject has a history of surgery within 3 months prior to administration, or failure to recover from surgery, or having an expected surgical plan during the trial;
6. Subject has abnormal vital signs, laboratory abnormalities, and ECGs;
7. Subject has used any of over-the-counter products within 7 days or prescription medications within 28 days prior to dosing;
8. Subject positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis seroreactivity (Trust);
9. Subject has a history of alcohol abuse within 1 year or positive alcohol breath test results;
10. Subject has a history of substance abuse within 1 year or a positive urine drug screen;
11. Subject who has daily smoking of ≥ 5 cigarettes within 3 months;
12. Subject who has special requirements for food, cannot comply with the unified diet or have dysphagia
13. Subject who has consumption of xanthine-rich foods or beverages (such as tea, coffee, cola, or chocolate) within 3 days prior to administration;
14. Subject who has consumption of food or beverages containing grapefruit within 7 days prior to administration;
15. Subject who has participated in other clinical trials and were enrolled/randomized within 3 months before administration;
16. Subject has used blood products or being blood donor or blood loss within 3 months;
17. Pregnant, lactating women, or positive pregnancy test;
18. Subject who refusal to contraception, or plan to donate sperm or ovums;
19. Other conditions which would make participation in the study unsuitable

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Predose and up to 240 hours postdose
Area Under the Curve from time 0 to the last measurable concentration (AUC0-t) | Predose and up to 240 hours postdose
Area Under the Curve from time 0 extrapolated to infinity (AUC0-inf) | Predose and up to 240 hours postdose

SECONDARY OUTCOMES:
Treatment-emergent adverse event | from baseline to day 25
Time to maximum concentration (Tmax) | Predose and up to 240 hours postdose
Half-life (t1/2) | Predose and up to 240 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Hufang Li, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No